CLINICAL TRIAL: NCT07028944
Title: Prospective Analysis of Medial Clear Space Widening in Weber B Ankle Fractures: A Comparison of Three Methods
Brief Title: Analysis of Medial Clear Space Widening in Weber B Ankle Fractures
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lucas Marchand, Principle Investigator, University of Utah
Other Study IDs: 162103
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Weber B Ankle Fractures
Keywords: Weber B ankle fractures; Medial Clear Space (MCS) Widening; gravity assisted stress (GAS); manual external rotation stress (MERS); weight-bearing stress (WBS); radiographs; X-rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Gravity assisted stress: Radiograph of ankle fracture under gravity assisted stress (7-10 days post-fracture, one-time clinic visit x-ray).
  Interventions: Other: Gravity assisted stress
- Manual external rotation stress: Radiograph of ankle fracture under manual external rotation stress (7-10 days post-fracture, one-time clinic visit x-ray, ).
  Interventions: Other: Manual external rotation stress
- Weight-bearing stress: Radiograph of ankle fracture under weight-bearing stress (7-10 days post-fracture, one-time clinic visit x-ray).
  Interventions: Other: Weight-bearing stress

INTERVENTIONS:
Other: Gravity assisted stress — Patients have a post 7-10 day ankle fracture x-ray taken under gravity assisted stress
  Groups: Gravity assisted stress
Other: Manual external rotation stress — Patients have a post 7-10 day ankle fracture x-ray taken under manual external rotation stress
  Groups: Manual external rotation stress
Other: Weight-bearing stress — Patients have a post 7-10 day ankle fracture x-ray taken under manual weigh-bearing stress
  Groups: Weight-bearing stress

SUMMARY:
The investigators purpose of this study is to obtain all three standard of care stress views of the ankle (gravity stress, manual stress, weightbearing stress) to compare the amount of tibiotalar joint instability predicted by each to determine if there are significant differences measured by the differing stress techniques.

DETAILED DESCRIPTION:
Rotational ankle injuries are a commonly encountered injury. Classification of these injuries is most commonly by the Danis-Weber (or Weber) classification and the Lauge-Hansen classification.

Within this classification system exists the isolated Weber B or Lauge-Hansen Supination External Rotation 2/4 (SER 2/4) injury which radiographically involves an isolated spiral fracture of the lateral malleolus at the level of the tibiofibular syndesmosis.

The difference between SER2 (isolated) Weber B injuries and SER4 injuries is disruption of the medial ankle mortise structures, either the medial malleolus (4a) or deltoid ligaments (4b) which then can permit increased talar subluxation with potential to result in tibitotalar joint incongruity.

Standard practice is to proceed with operative fixation of rotationally unstable Weber B or SER4b injuries.

To determine the competence of medial ligamentous structures in isolated fractures of the fibula at the level of the syndesmosis when there is minimal widening of the mortise on non weight bearing films there are three plain x-ray views currently widely used and considered standard of care:

1. manual external rotation stress;
2. gravity assisted stress;
3. and weight-bearing stress radiographs.

Increased widening on one of these views is used to decide whether to treat the fracture with or without surgery.

Globally there is wide variability as to which stress-view radiograph or combination of these are used. To our knowledge, no study to date has compared all three stress-view radiographs concurrently to determine if the three different methods predict equal amounts of tibiotalar joint instability.

The need to understand how these three views compare is crucial, as tibiotalar instability is primary indication for surgical stabilization.

The null hypothesis therefore is the investigators will find no difference in the tibiotalar joint instability between the three stress views.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Weber B ankle fracture who are skeletally mature (no open physes) and older than 18 years of age.

Exclusion Criteria:

* Medial and/or posterior Malleolar fracture
* Any other lower extremity trauma that limits weight bearing
* Concomitant arthridities/rheumatologic disease (patients with osteoarthritis may be included)
* Prior fracture
* Prior surgery of foot, talus or ankle
* Open fracture
* Initial NWB xrays with a medial clear space (MCS) > 7 mm or medial clear space> superior clear space (SCS) by 2mm, signifying an unstable fracture prior to stress
* Protected populations

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age with a Weber B ankle fracture who are skeletally mature (no open physes).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Medial Clear Space (MCS) Widening Under Gravity Assisted Stress | Day 1 Clinic Visit
  Measured distance, millimeters(mm) of the fractured fibula at the level of the syndesmosis joint in patients undergoing gravity assisted stress
Medial Clear Space (MCS) Widening Under Manual External Rotation Stress | Day 1 Clinic Visit
  Measured distance, millimeters(mm) of the fractured fibula at the level of the syndesmosis joint in patients undergoing manual external rotation stress
Medial Clear Space (MCS) Widening Under Weight-bearing Stress | Day 1 Clinic Visit
  Measured distance, millimeters(mm) of the fractured fibula at the level of the syndesmosis joint in patients undergoing weight-bearing stress

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Marchand, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States